CLINICAL TRIAL: NCT04334395
Title: A Retrospective Cohort Study Outcome of Treatment in Asymptomatic Stage 4 Colorectal Cancer : Primary Tumor Resection vs. No Primary Tumor Resection
Brief Title: A Retrospective Cohort Study Outcome of Treatment in Asymptomatic Stage 4 Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: MURA2016/546
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Stage IV Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: primary tumor resection group — resection of cancer at colon

SUMMARY:
In asymptomatic Stage 4 colorectal cancer, the treatment varies between many hospitals and countries. Some studies found that primary tumor resection had better survival rates and a lower risk of mortality. But many studies found significant benefits in survival in sub groups of the population such as age less than 70 years, WHO performance status <2, no extra-hepatic metastasis, liver tumor burden <50%. However some studies showed no survival benefits in primary tumor resection. So this study will focus on survival, adverse events, complications in primary tumor resection and no primary tumor resection in asymptomatic Stage 4 colorectal cancer.

DETAILED DESCRIPTION:
The retrospective study of patients in asymptomatic Stage 4 colorectal cancer received treatment at Ramathibodi Hospital and excluded symptomatic primary tumors such as obstruction, perforation that required surgery, carcinomatosis peritoneii, and patients with secondary cancer diagnosis in the past 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic stage IV colorectal cancer
* pathological prove adenocarcinoma
* age >18 years
* no primary tumor related symptom
* ECOG performance status <2

Exclusion Criteria:

* symptomatic primary tumor such as obstruction , perforation that required surgery
* carcinomatosis peritoneii
* patients with secondary cancer diagnosis in 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medical records of stage IV colorectal cancer with unresectable distant metastasis received treatment in Ramathibodi hospital between 1 September 2006 - 31 August 2016.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Complication rate | 5 year
  The definition of complication defined as symptom that occurred during treatment period such as obstruction , perforation , bleeding , trenesmus.

SECONDARY OUTCOMES:
The survival time | 5 year
  The survival time defined as time from diagnosis to death or last follow up period

CONTACTS AND LOCATIONS:
Overall Officials: Chairat Supsamutchai, MD, Study Chair — 270, Rama VI road, Ratchathevi, Deapartment of Surgery, Faculty of Medicine, Ramathibodi Hospital, Mahidol University, Bangkok, Thailand, 10400
Locations (1):
- Chairat Supsamutchai, Bangkok, Bankok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided